CLINICAL TRIAL: NCT03830411
Title: A Phase II, Prospective, Single-center, Randomized, Controlled Study to Investigate the Efficacy and Safety of Sintilimab Compared With Docetaxel or Pemetrexed as Second-line Treatment for Patients With Stage IV Nonsquamous Non-small Cell Lung Cancer With Wild-type EGFR After Failure With Platinum-Containing Chemotherapy.
Brief Title: A Study of Sintilimab Compared With Docetaxel or Pemetrexed as Second-line Treatment for Patients With Stage IV Nonsquamous Non-small Cell Lung Cancer After Failure With Platinum-Containing Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xin-Hua Xu (Other)
Responsible Party: Sponsor-Investigator, Xin-Hua Xu, professor, China Three Gorges University, Yichang, China
Organization: China Three Gorges University, Yichang, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTGU002
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Nonsquamous Non-Small Cell Lung Cancer
Keywords: Sintilimab; docetaxel; pemetrexed; nonsquamous non-small-cell lung cancer; wild-type EGFR; second-line treatment
MeSH Terms: interventions — sintilimab; Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Sintilimab (Experimental): Participants will receive Sintilimab as long as they continue to experience clinical benefit in the opinion of the investigator until unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator.
  Interventions: Drug: Sintilimab
- Arm B: Chemotherapy (Docetaxel or Pemetrexed) (Active Comparator): Participants randomized to the chemotherapy arm will receive docetaxel or pemetrexed until disease progression per standard RECIST v1.1 or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: Sintilimab — Sintilimab will be administered intravenously at a fixed dose of 200 milligrams (mg) on Day 1 of each 21-day cycle.
  Other Names: IBI308
  Arms: Arm A: Sintilimab
Drug: Docetaxel — Docetaxel 75 milligrams per square meter (mg/m^2) will be administered intravenously on Day 1 of each 21-day cycle.
  Arms: Arm B: Chemotherapy (Docetaxel or Pemetrexed)
Drug: Pemetrexed — Pemetrexed 500 mg/m^2 will be administered intravenously on Day 1 of each 21-day cycle.
  Arms: Arm B: Chemotherapy (Docetaxel or Pemetrexed)

SUMMARY:
This prospective, single-center, randomized, controlled study will evaluate the efficacy and safety of sintilimab compared with docetaxel or pemetrexed as second-line treatment for patients with stage IV nonsquamous non-small cell lung cancer with wild-type EGFR after failure with platinum-containing chemotherapy. Treatment may continue as long as participants are experiencing clinical benefit as assessed by the investigator, i.e., in the absence of unacceptable toxicity or symptomatic deterioration attributed to disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research; fully understand and know the research and sign informed consent;
2. Age ≥ 18 years old and ≤ 75 years old, either sex;
3. Eastern Collaborative Oncology Group Performance status (ECOG PS) 0, 1 or 2;
4. Has a histologically or cytologically confirmed diagnosis of stage IV (according to the 8th edition of the International Association for the Study of Lung Cancer) nonsquamous NSCLC;
5. Have at least one measurable lesion as defined by RECIST 1.1;
6. Has progression of disease after treatment with at least two cycles of a platinum-containing doublet chemotherapy according to RECIST V.1.1;
7. Patients without activating EGFR mutation;
8. Normal hepatic function: total bilirubin≤1.5×normal upper limit (ULN); Alanine aminotransferase and Aspartate aminotransferase levels ≤2.5×ULN or ≤5×ULN if liver metastasis is present;
9. Normal renal function: Creatinine ≤1.5×ULN or calculated creatinine clearance ≥45 mL/min (using Cockcroft/Gault formula to calculate );
10. Normal hematological function: absolute neutrophil count ≥1.5×109/L, platelet count ≥70×109/L, hemoglobin≥80g/L [no blood transfusion or erythropoietin (EPO) within 7 days] Dependency];
11. Has a life expectancy of at ≥3 months.

Exclusion Criteria:

1. ECOG PS >2;
2. Small cell lung cancer and squamous NSCLC;
3. EGFR mutation or mutation status unknown;
4. Known hypersensitivity or allergy to monoclonal antibody;
5. Prior therapy with an anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2, anti-tumor necrosis factor CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways);
6. Active autoimmune disease, or a documented history of autoimmune disease;
7. Treatment with systemic corticosteroids (prednisone≥10mg per day or equivalent dose) or other systemic immunosuppressive medications within 2 weeks prior to the first dose;
8. Known history or active human immunodeficiency virus (HIV);
9. Known acute or chronic active hepatitis B (HBV DNA positive) infection or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive) infection;
10. Interstitial lung disease, or history of pneumonitis requiring systemic steroids for treatment;
11. Active or poorly controlled severe infection;
12. Have serious cardiovascular disease: Symptomatic congestive heart failure (New York Heart Association grade III-IV), unstable angina pectoris, unstable arrhythmia, myocardial infarction or cerebrovascular accident within 3 months before randomization;
13. Received thoracic radiation therapy of >30 Gy within 6 months prior to first dose of study drug;
14. Completed palliative radiotherapy within 7 days prior to first dose of study drug;
15. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Approximately 21 months
  Overall Survival (OS) was defined as the time from the date of randomization to the date of death due to any cause. Data for participants who were not reported as dead at the time of analysis was censored at the date when they were last known to be alive.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 21 months
  ORR was defined as the percentage of participants with confirmed objective tumor response, complete response (CR) or partial response (PR), as determined by investigator using RECIST v1.1 criteria.
Progression-free survival (PFS) | Approximately 21 months
  PFS was defined as the time between the date of randomization and the date of first documented disease progression or death, whichever occurs first. Disease progression was determined based on investigator assessment using response evaluation criteria In solid tumors (RECIST) v1.1.
Duration of response (DOR) | Approximately 21 months
  DOR was defined as the duration from the first tumor assessment that supports the participant's objective response (CR or PR, whichever is first recorded) to disease progression or death due to any cause, whichever occurs first.
Emergence of adverse events(AEs) | Approximately 21 months
  AEs graded using CTCAE (Version 4.0) criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Central Hospital of Yichang City, the First Clinical Medical College of Three Gorges University, Yichang, Hubei, China

IPD SHARING:
Plan to Share IPD: No